CLINICAL TRIAL: NCT03048461
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial Investigating the Effect of Autologous Platelet-rich Plasma in Subjects With Androgenetic Alopecia.
Brief Title: The Effect of Platelet-rich Plasma in Subjects With Androgenetic Alopecia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not want to enroll and proceed with this study concept.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, MD, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA04222016
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Platelet Rich Plasma (Experimental): Participants will receive intradermal injections autologous PRP to an area (100cm2) of alopecia on the scalp.Two treatments will be performed 3 months apart
  Interventions: Device: Platelet Rich Plasma Prep System
- Placebo (sterile saline) (Placebo Comparator): Participants will receive intradermal injections of sterile normal saline to an area (100cm2) of alopecia on the scalp. Two treatments will be performed 3 months apart
  Interventions: Device: Platelet Rich Plasma Prep System; Drug: Placebo

INTERVENTIONS:
Device: Platelet Rich Plasma Prep System — intradermal injections of platelet rich plasma to an area of alopecia
Drug: Placebo — intradermal injections to an area of alopecia
  Arms: Placebo (sterile saline)

SUMMARY:
The purpose of this study is to evaluate the effect of autologous platelet-rich plasma (PRP) in the treatment of androgenetic alopecia.

This is a randomized clinical trial to evaluate the effect of autologous platelet rich plasma in subjects with moderate androgenetic alopecia. Approximately 30 subjects will be randomized into the study. The study is designed as an 18-month study consisting of 2 phases. This study was a pilot study designed to determine feasibility of this procedure.

Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years old and ≤55 years old
2. Subjects are in good health as judged by the investigator.
3. Diagnosed with by a dermatologist with moderate androgenetic alopecia.
4. Subject is seeking treatment for androgenetic alopecia.
5. Subject has never previously used finasteride or minoxidil or has consistently used finasteride or minoxidil for at least 1 year.
6. Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.

Exclusion Criteria:

1. Other than androgenetic alopecia, evidence of another skin condition affecting the treatment area that would interfere with clinical assessments.
2. Subjects who are unwilling to avoid initiating treatment with minoxidil or finasteride for the duration of the study; or in subjects who have been treated with minoxidil or finasteride for at least 1 year, unwilling to avoid changes in the dosing regimen of these medications for the duration of the study.
3. Willing to refrain from washing hair or using hair product 24 hours before and after treatment visits
4. History of a clinically significant hematologic disorder as determined by the investigator.
5. Subjects currently receiving anticoagulant or anti-platelet therapy.
6. Subjects on daily Aspirin therapy for cardiovascular disease.
7. Subjects with chronic NSAID use, unable to wean off.
8. Subject is known to be HIV positive.
9. History of recurrent facial or labial herpes simplex infection
10. History of hypertrophic scars or keloids
11. Known genetic disorders affecting fibroblasts or collagen, such as achondroplasia, osteogenesis imperfecta, etc.
12. Subjects who have any requirement for the use of local or systemic steroids or other immunosuppressive agent
13. Pregnant or breast feeding
14. Uncooperative patients or patients with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.
15. Subjects who are unable to understand the protocol or give informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Clinical change of androgenetic alopecia, as determined by scoring photographs | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University